CLINICAL TRIAL: NCT00398554
Title: Pilot Study for Therapy Optimising for Hodgkin's Lymphoma in Childhood and Adolescence; Optimising Therapy for Boys With Hodgkin's Lymphoma in Intermediate and Advanced Stages. Safety and Efficacy Study for Drug Combination VECOPA
Brief Title: Combination Chemotherapy in Treating Young Male Patients With Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christine Mauz-Körholz (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Sponsor-Investigator, Christine Mauz-Körholz, Study Secretary of the EuroNet-PHL group, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000514344; GPOH-HD-2002-PILOT-VECOPA; EU-20652; EUDRACT-2004-005244-28
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vinblastine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VECOPA (Experimental): dose and time intensified consoloditation chemotherapy cycle
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vinblastine sulfate; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — 1250 mg/m2 i.v. 60 Min.-Inf. day 1 and 21
Drug: doxorubicin hydrochloride — 25mg/m²/day, 2 hours i.v.infusion on day 21
Drug: etoposide — 150 mg/m²/day, 2 hours i.v.infusion (intravenous drip) on days 1 - 3
Drug: prednisone — 40 mg/m2/day p.o. (intake by mouth)divided in 3 single doses daily from day 1 - 14 and day 21 - 34
Drug: vinblastine sulfate — 6 mg/m² i.v. bolus on day 1 and day 21
Drug: vincristine sulfate — 1,5 mg/m2 i.v. bolus max. single dose 2 mg (cap dose at 2 mg) on day 8 and day 29
Radiation: radiation therapy — involved field irradiation, single daily fractions 1,5 Gy to max. 1,8 Gy standard dose 20 Gy, max dose 30 Gy (boost irradiation if required)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well combination chemotherapy works in treating young male patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of combination chemotherapy comprising vincristine, etoposide, cyclophosphamide, vinblastine, prednisone, and doxorubicin hydrochloride (VECOPA) in pediatric male patients with previously untreated stage II-IV classic Hodgkin's lymphoma.
* Compare the effects of VECOPA vs cyclophosphamide, vincristine, procarbazine hydrochloride, and prednisone (COPP) in these patients.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to disease stage (IA/B[E], IIA[E], IIB, or IIIA vs IIB[E], IIIA/B[E], IIIB, or IVA/B).

* Stratum 1 (stages IA/B[E], IIA[E], IIB, or IIIA): Patients receive oral prednisone on days 1-15, vincristine IV on days 1, 8, and 15, doxorubicin hydrochloride IV over 4 hours on days 1 and 15, and etoposide IV over 2 hours on days 2-6 (OEPA). Treatment repeats every 4 weeks for 2 courses. Beginning at week 9, patients receive VECOPA chemotherapy comprising oral prednisone on days 1-14 and 21-34, etoposide IV over 2 hours on days 1-3, doxorubicin hydrochloride IV over 2 hours on day 21, vinblastine IV and cyclophosphamide IV over 1 hour on days 1 and 21, and vincristine IV on days 8 and 29. Patients then undergo radiotherapy.
* Stratum 2 (stages IIB[E], IIIA/B[E], IIIB, or IVA/B): Patients receive 2 courses of OEPA as in stratum 1 followed by 2 courses of VECOPA (6-week courses). Patients then undergo radiotherapy.

After completion of study treatment, patients are followed periodically for at least 6 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of classic Hodgkin's lymphoma (HL)

  * Intermediate or advanced disease (stage I[E]-IV)
* No lymphocyte-predominant HL
* Previously untreated disease

PATIENT CHARACTERISTICS:

* Male
* No known hypersensitivity or contraindication to study drugs
* No other concurrent malignancies
* No severe concurrent diseases (e.g., immune deficiency syndrome)
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy
* More than 30 days since prior and no other concurrent investigational drugs
* More than 30 days since prior and no concurrent participation in another clinical trial

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2005-06; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Toxicity at days 21 and 42 (+/- 2 days) of treatment | days 21 and 42 (+/- 2 days) of treatment after start of VECOPA cycle
  number of VECOPA cycles that allow continuation of chemotherapy on a sufficient hematopoietic recovery

SECONDARY OUTCOMES:
Event-free survival | event-free survival at 5 years
Overall survival | overall survival at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koerholz, MD, Study Chair — Martin-Luther-Universität Halle-Wittenberg
Locations (12):
- Germany (11):
  - Klinikum Augsburg, Augsburg
  - Charite University Medical Center of Berlin, Berlin
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsfrauenklinik Frankfurt, Frankfurt
  - Universitaetsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets - Kinderklinik, Leipzig
  - Kinderklinik d. TU / Schwabing, Munich
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Klinikum Oldenburg, Oldenburg
- University Children's Hospital, Zurich, Switzerland